CLINICAL TRIAL: NCT05648357
Title: A Single-arm, Open-label, Multi-center, Phase IV Trial to Evaluate the Reactogenicity, Safety, and Immunogenicity of Quadrivalent Seasonal Influenza Vaccine (Fluarix Tetra) in Participants Aged 65 Years and Older in India
Brief Title: A Study to Assess the Safety and Immune Response of Quadrivalent Seasonal Influenza Vaccine (Fluarix Tetra) in Participants Aged 65 Years and Older in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 218702
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quadrivalent seasonal influenza (FLU D-QIV) vaccine group (Experimental): Participants received 1 dose of seasonal FLU vaccine at Day 1.
  Interventions: Biological: Fluarix Tetra Vaccine

INTERVENTIONS:
Biological: Fluarix Tetra Vaccine — A single dose of Fluarix Tetra vaccine administered intramuscularly (IM) on day 1.

SUMMARY:
The purpose of this study is to gather additional evidence of the safety and immunogenicity of 1 dose of Fluarix Tetra (0.5 milliliter [mL]) (Northern Hemisphere (NH)2023-2024) in individuals aged 65 years and above to fulfill a post-approval condition imposed by the Indian regulatory authorities (CDSCO) for this age group in India.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged >= 65 years of age
* Participants and/or legally acceptable representative (s) (LAR) who in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits
* Written or witnessed/thumb printed informed consent obtained from the participant and/or participant's LAR(s) after the study has been explained according to the local authority requirements and prior to performance of any study-specific procedure

Exclusion Criteria:

* History of severe allergic reactions (e.g., anaphylaxis) to any component of the vaccine, including egg protein, or following a previous dose of any influenza vaccine.
* Receipt of licensed vaccine, immune sera and/or any blood products, or an investigational trial agent within previous 30 days or planned during their participation in the trial.
* Receipt of any flu vaccine within 6 months before trial start or any other vaccine within 30 days before the trial.
* Receipt of any dose of a Coronavirus Disease 2019 (COVID-19) vaccine within 15 days of trial start.
* History of Guillain-Barré Syndrome.
* Altered immune status or chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying agents within six months prior to administration of trial vaccine.
* History of acute infectious disease or acute respiratory illness needing antibiotics or antivirals in the previous 7 days, based on investigator's judgement.
* If a participant candidate has fever, the trial vaccination should be postponed to when the fever has resolved for at least 2 days (temporary exclusion criterion). Fever is defined as temperature >=38.0 degree Celsius (°C) (100.4 degrees Fahrenheit [°F]) by any route. The preferred location for measuring temperature will be oral route.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by medical history, physical examination, or laboratory screening tests.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- India (5):
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Kattankulathur
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Varanasi
  - GSK Investigational Site, Visakhapatnam

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Jain V, Cauwberghs F, Qian H, Best-Sule K, Gupta V, Tatchou EN, Struyf F. Reactogenicity, safety, and immunogenicity of a quadrivalent seasonal influenza vaccine in adults aged 65 years and older: Phase 4 study results from India during December 2023-February 2024. Hum Vaccin Immunother. 2025 Dec;21(1):2578084. doi: 10.1080/21645515.2025.2578084. Epub 2025 Oct 29. PMID 41159757

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Started | 250
Completed | 247
Not Completed | 3
Not completed — CONSENT WITHDRAWAL, NOT DUE TO AN AE | 3

BASELINE CHARACTERISTICS:
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 250
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 71.8 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 146
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central / South Asian Heritage | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Adverse Event
Description: The solicited administration site adverse events included pain, redness and swelling.
Time Frame: Day 1 to Day 7
Population: The analysis was performed on the Solicited Safety Set (SSS), which included participants that received study intervention and had solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 247
Participants | 44

2. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: The solicited systemic events included fever, headache, myalgia (muscle pain), arthralgia (joint pain), fatigue, gastrointestinal symptoms (including nausea, vomiting, diarrhea and/or abdominal pain), sweating and shivering.
Time Frame: Day 1 to Day 7
Population: SSS population
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 247
Participants | 30

3. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is defined as an event reported in addition to the solicited AEs during the clinical study. Also, any solicited symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event.
Time Frame: Day 1 to Day 21
Population: Analysis was performed on Exposed Set (ES) population, which included all participants that received the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 250
Participants | 4

4. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: A SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: Day 1 to Day 21
Population: ES population
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 250
Participants | 0

5. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination-inhibiting (HI) Antibodies
Description: Serum HI antibodies against the four-influenza vaccine strains are expressed as GMTs, in titers. The assessed strains are: A/Victoria/4897/2022 (H1N1), A/Darwin/9/2021 (H3N2), B/Austria/1359417/2021 and B/Phuket/3073/2013.
Time Frame: At Baseline (Day 1) and Day 22
Population: Analysis was performed on the Per Protocol Set (PPS), which included all participants who received the trial intervention as per protocol, had immunogenicity results pre- and post-dose, complied with the allowed dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 211
Titer
  A/Victoria/4897/2022 (H1N1), Day 1 | 10.7 [9.2 to 12.4]
  A/Victoria/4897/2022 (H1N1), Day 22 | 187.9 [150.2 to 235.1]
  A/Darwin/9/2021 (H3N2), Day 1 | 20.2 [17.0 to 23.9]
  A/Darwin/9/2021 (H3N2), Day 22 | 205.3 [169.5 to 248.8]
  B/Austria/1359417/2021, Day 1 | 100.8 [87.8 to 115.9]
  B/Austria/1359417/2021, Day 22 | 903.6 [780.4 to 1046.3]
  B/Phuket/3073/2013, Day 1 | 93.3 [82.0 to 106.2]
  B/Phuket/3073/2013, Day 22 | 701.6 [611.7 to 804.7]

6. Secondary Outcome: Mean Geometric Increase (MGI) of Serum HI Antibodies
Description: MGI is defined as the fold increase in post-vaccination serum HI GMTs compared with Baseline. Analysis was performed for four influenza strains: A/Victoria/4897/2022 (H1N1), A/Darwin/9/2021 (H3N2), B/Austria/1359417/2021 and B/Phuket/3073/2013.
Time Frame: At Day 22 (compared with Baseline [Day 1])
Population: PPS population
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 211
Fold increase
  A/Victoria/4897/2022 (H1N1) | 17.6 [13.6 to 22.9]
  A/Darwin/9/2021 (H3N2) | 10.2 [8.2 to 12.7]
  B/Austria/1359417/2021 | 9.0 [7.5 to 10.7]
  B/Phuket/3073/2013 | 7.5 [6.4 to 8.9]

7. Secondary Outcome: Number of Participants With Seroconversion Rate (SCR)
Description: SCR is defined as the percentage of participants who have either a pre-vaccination titer less than (<) 1:10 and a postvaccination titer greater than or equal to (>=) 1:40 or a pre-vaccination titer >= 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 22
Population: PPS population
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 211
Participants
  A/Victoria/4897/2022 (H1N1) | 169
  A/Darwin/9/2021 (H3N2) | 160
  B/Austria/1359417/2021 | 173
  B/Phuket/3073/2013 | 162

8. Secondary Outcome: Number of Participants With Seroprotection Rate (SPR)
Description: SPR is defined as the percentage of participants with a serum HI titer >=1:40.
Time Frame: At Day 1 and Day 22
Population: PPS population
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
Number analyzed (Participants) | 211
Participants
  A/Victoria/4897/2022 (H1N1), Day 1 | 40
  A/Victoria/4897/2022 (H1N1), Day 22 | 180
  A/Darwin/9/2021 (H3N2), Day 1 | 69
  A/Darwin/9/2021 (H3N2), Day 22 | 187
  B/Austria/1359417/2021, Day 1 | 182
  B/Austria/1359417/2021, Day 22 | 209
  B/Phuket/3073/2013, Day 1 | 186
  B/Phuket/3073/2013, Day 22 | 210

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during a 7-day period after vaccine administration (from Day 1 to Day 7). Unsolicited AEs and SAEs were collected during a 21-day period after vaccine administration (from Day 1 to Day 21).
Arm/Group | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 70/250
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Seasonal Influenza (FLU D-QIV) Vaccine Group (N=250)
Administration site erythema (General disorders) | 5 (5)
Administration site pain (General disorders) | 37 (37)
Administration site swelling (General disorders) | 4 (4)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 16 (16)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pustule (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9)
Headache (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05648357/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT05648357/SAP_001.pdf